CLINICAL TRIAL: NCT05385666
Title: Collaborative Mental Health Care Model: an Evaluation of the Implementation of a Pilot in Four Health Homes
Brief Title: Collaborative Mental Health Care Model: an Evaluation of the Implementation of a Pilot in Four Primary Care Organization
Acronym: Mosaique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Nadia YOUNES (Other)
Responsible Party: Sponsor-Investigator, Dr Nadia YOUNES, Investigator Coordinator, Versailles Hospital
Organization: Versailles Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: P21/10_mosaïque
Record Dates: First submitted 2022-05-12; First posted 2022-05-23 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Psychological Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group experimental (Experimental)
  Interventions: Other: collaborative cares

INTERVENTIONS:
Other: collaborative cares — coordinate care between city medicine and specialized psychiatric care to improve the management of common mental disorders

SUMMARY:
Frequent mental disorders (anxiety or mood disorders), an important part of primary care patient care, remain insufficiently detected and treated. Improving their care requires better coordination between general practice and specialized care. The collaborative care model developed in Washington State with the introduction of a care manager is recognized. About 100 randomized controlled trials have established its effectiveness and efficiency, in terms of improving the progression of disorders (remission rate), adherence, quality of life, professional and patient satisfaction, and cost savings. However, the possibility of implementation of these validated care remains to be explored. A dozen collaborative care implementation studies exist, all conducted in the USA and not having considered all the dimensions of the indicators of penetration, acceptability/adoption, feasibility, fidelity and cost. A first implementation in France is implemented since September 2021 in the Yvelines department on four sites of different size, organization and environments: the multi-professional health centers (MSP) of Mureaux and Celle St Cloud, the Chevreuse medical house and MG in isolated practice in Versailles.

The main objective of the research project is to evaluate the first implementation in France of collaborative care for frequent psychic disorders according to the indicators of penetration, acceptability/adoption, fidelity, relevance, feasibility and cost.

ELIGIBILITY:
Inclusion Criteria:

* healthcare professionals involved in the collaborative care system
* patients who have been referred for collaborative care by their family physician

Exclusion Criteria:

* patient refusal to participate in research
* adults protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
to evaluate the first implementation in France of collaborative care for frequent psychic disorders | 36 months
  numbers of patients and medical caregivers who participate in collaborative care

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Maison de Santé Pluridisciplinaire, Chevreuse
  - Maison de Santé Pluridisciplinaire, Les Mureaux
  - Cabinet Médical Versailles, Versailles
  - cabinet médical Versailles, Versailles

IPD SHARING:
Plan to Share IPD: Undecided